CLINICAL TRIAL: NCT01757821
Title: 6-Hz Primed vs. Unprimed Low-Frequency rTMS in Chronic Stroke
Brief Title: Primed vs. Unprimed rTMS in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BrainPrime
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Stroke
Keywords: Stroke; rTMS; TMS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 6-Hz Priming (Experimental): real 6-Hz primed low-frequency rTMS
  Interventions: Device: real 6-Hz primed low-frequency rTMS
- Sham 6-Hz Priming (Sham Comparator): Sham 6-Hz Primed low-frequency rTMS
  Interventions: Device: Sham 6-Hz Primed low-frequency rTMS
- Real 1-Hz rTMS only (Active Comparator): real 1-Hz rTMS only
  Interventions: Device: real 1-Hz rTMS only

INTERVENTIONS:
Device: real 6-Hz primed low-frequency rTMS — 10 minutes of 6-Hz stimulation (real priming) followed by 10 minutes of 1-Hz low-frequency stimulation delivered to the nonstroke primary motor region
  Arms: 6-Hz Priming
Device: Sham 6-Hz Primed low-frequency rTMS — 10 minutes of sham priming stimulation followed by 10 minutes of 1-Hz low-frequency stimulation delivered to the nonstroke primary motor region
  Arms: Sham 6-Hz Priming
Device: real 1-Hz rTMS only — 20 minutes of low-frequency rTMS delivered to the nonstroke primary motor region
  Arms: Real 1-Hz rTMS only

SUMMARY:
The goal of stroke rehabilitation is to restore function to the weak side of the body. However, this is often a difficult task to accomplish due to not only to damage from the stroke, but from increased excitability in the non-stroke side of the brain that inhibits the stroke side from functioning optimally. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive form of brain stimulation that can enhance excitability in the stroke side when applied at a low-frequency on the non-stroke side. By "inhibiting the inhibition" (i.e. disinhibition), rTMS promotes adaptive brain reorganization following stroke. Previous research in healthy individuals demonstrates enhanced effects of low-frequency rTMS when it is preceded by high-frequency (excitatory) rTMS stimulation known as priming. Our lab previously demonstrated the safety of 6-Hz priming with low-frequency rTMS in both adults and children with chronic stroke. However, it is currently unknown whether or not the addition of priming stimulation to low-frequency rTMS enhances excitability in the stroke hemisphere. Our study will examine three rTMS interventions in twelve adults (at least 18 years): 1.) 10 minutes of real priming followed by 10 minutes of low-frequency rTMS, 2.) 10 minutes of fake priming followed by 10 minutes of low-frequency rTMS, 3.) 20 minutes of low-frequency rTMS only. Participants will receive all three interventions in randomized order. Each week, participants will complete two pretest and 3 posttest sessions consisting of behavioral measures of weak upper extremity function and cortical excitability in addition to receiving one rTMS intervention. Following each week of testing and treatment, subjects will take a one week rest break before crossing-over to receive another intervention. We hypothesize the following: 1.) Primed rTMS will result in significantly reduced inhibition and significantly increased excitation on the stroke side vs. fake primed rTMS or low-frequency rTMS given alone and 2.) Primed rTMS will result in greater improvements of paretic hand function. This study is innovative in that it intends to compare primed and unprimed rTMS in the stroke brain that could acknowledge a more effective delivery method of rTMS to potentially yield greater rehabilitative outcomes.

DETAILED DESCRIPTION:
Recovery following stroke is difficult not only because of the neuronal death from the ischemic insult but also because of maladaptive brain reorganization occurring from exaggerated inhibition imparted by the over-compensating contralesional primary motor area (M1) onto the ipsilesional M1 via transcallosal pathways. Advancement in stroke rehabilitation depends on innovative treatments like repetitive transcranial magnetic stimulation (rTMS) that possess the ability to disrupt this excessive inhibition. Through previous NIH/NICHD funding, my sponsor's research team confirmed the safety and efficacy of rTMS in both adult (1R01 HD053153-01A2) and children (1RC1 HD063838-01) with stroke using 6-Hz primed low-frequency rTMS applied to the contralesional M1 to produce disinhibition of the ipsilesional M1. With feasibility of primed rTMS now demonstrated, the proposed research plan will directly compare primed rTMS to unprimed rTMS. The investigators will investigate whether pretreatment of inhibitory low-frequency rTMS with excitatory high-frequency priming is more effective than sham-primed low-frequency rTMS in correcting the exaggerated interhemispheric inhibition acting on ipsilesional M1. While this may sound contradictory, the Bienenstock-Cooper-Munro theory of bidirectional plasticity supports this concept. The long-term goal is to discover the most effective rTMS protocol with which to safely up-regulate ipsilesional M1, rendering a more potent neuronal network for voluntary recruitment. By studying the efficacy of priming as measured by the amount of cortical excitability in both ipsilesional and contralesional hemispheres, a more advantageous delivery of rTMS may be realized and eventually incorporated into research trials and clinical practice. The study poses significant innovation as it explores the role of metaplasticity in rehabilitation using rTMS. The investigators will employ a double-blind crossover study using twelve adult participants with stroke. Because of heterogeneity in stroke type and location between subjects, a crossover design will reduce variability as each subject serves as their own control.

Specific Aim #1: Compare the effect of 6-Hz primed vs. unprimed low-frequency rTMS on cortical excitability in chronic stroke.Cortical excitability will be explored with TMS using ipsilesional paired-pulse testing, cortical silent period testing, and interhemispheric inhibition (IHI) paired-pulse testing.

Working hypotheses are:

1. Primed rTMS will result in greater increases in the 3-ms and 15-ms ipsilesional paired-pulse to single-pulse (ipsilesional PP/SP) ratios than unprimed rTMS, indicating of decreased intracortical inhibition (GABAA-mediated) and greater intracortical facilitation, respectively.
2. Primed rTMS will result in greater decreases than unprimed rTMS in duration of cortical silent period, indicating decreased inhibition (GABAB-mediated).
3. Primed rTMS will result in a greater increase in the IHI PP/SP ratio in the non-stroke to stroke hemisphere direction and a corresponding decrease in the IHI PP/SP ratio in the stroke to non-stroke hemisphere direction than unprimed rTMS. This is consistent with less inhibition imparted onto the stroke hemisphere from the non-stroke hemisphere and greater inhibition imparted on the non-stroke hemisphere from the stroke hemisphere.

Specific Aim #2: Compare the effect of 6-Hz primed vs. unprimed low-frequency rTMS on functional outcome in chronic stroke. Functional outcome will be assessed by paretic hand performance on the Box and Block test.

Working hypothesis is:

1. Primed rTMS will result in greater improvements on the Box and Block test.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* presence of stroke at least six months duration
* demonstrate at least 10 degrees of active extension at the paretic index finger (metacarpophalangeal joint)
* possess resting motor evoked potential on the stroke hemisphere with TMS testing
* Upper Extremity Fugl Meyer score at least 20 out of 66
* Beck Depression Inventory equal to or less than 19 out of 63
* Mini-Mental State Examination score at least 24 out of 30
* age-appropriate receptive language ability

Exclusion Criteria:

* history of seizure within the last two years
* indwelling metal or medical devices incompatible with TMS
* anosognosia
* pregnancy
* any co-morbidities impairing upper extremity function (e.g. fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Carey, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects received all 3 interventions
Groups:
- 6-Hz Priming: real 6-Hz primed low-frequency rTMS
  real 6-Hz primed low-frequency rTMS: 10 minutes of 6-Hz stimulation (real priming) followed by 10 minutes of 1-Hz low-frequency stimulation delivered to the nonstroke primary motor region
  Sham 6-Hz Primed low-frequency rTMS
  real 1-Hz rTMS only
  real 1-Hz rTMS only: 20 minutes of low-frequency rTMS delivered to the nonstroke primary motor region
  Sham 6-Hz Primed low-frequency rTMS: 10 minutes of sham priming stimulation followed by 10 minutes of 1-Hz low-frequency stimulation delivered to the nonstroke primary motor region
Period: Overall Study
Arm/Group | 6-Hz Priming
Started | 11 (11 subjects)
Completed | 10 (10 subjects)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Real 6-Hz Priming Sham 6-Hz Priming Real 1-Hz rTMS Only: real 6-Hz primed low-frequency rTMS
  real 6-Hz primed low-frequency rTMS:
  Sham 6-Hz Primed low-frequency rTMS
  real 1-Hz rTMS only
Arm/Group | Real 6-Hz Priming Sham 6-Hz Priming Real 1-Hz rTMS Only
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Cortical Excitability: Paired-Pulse
Description: Cortical Excitability of the primary motor cortex on the stroke hemisphere will be assessed using paired-pulse transcranial magnetic stimulation.
Time Frame: Change from Baseline to 20 minutes
Measure: Mean (Standard Deviation); unit: milivolt
Groups:
- Real 6-Hz Priming: real 6-Hz primed low-frequency rTMS
  real 6-Hz primed low-frequency rTMS: 10 minutes of 6-Hz stimulation (real priming) followed by 10 minutes of 1-Hz low-frequency stimulation delivered to the nonstroke primary motor region
Arm/Group | Real 6-Hz Priming | Sham 6-Hz Priming | Real 1-Hz rTMS Only
Number analyzed (Participants) | 10 | 10 | 10
milivolt | -18 (14) | 18 (9) | 12 (5)

ADVERSE EVENTS:
Arm/Group | Real 6-Hz Priming | Sham 6-Hz Priming | Real 1-Hz rTMS Only
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/11 | 1/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real 6-Hz Priming (N=11) | Sham 6-Hz Priming (N=11) | Real 1-Hz rTMS Only (N=11)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No